CLINICAL TRIAL: NCT03334955
Title: Effect of Laparoscopic Ovarian Drilling on Subendometrial Blood Flow in Women With Polycystic Ovary Syndrome
Brief Title: Laparoscopic Ovarian Drilling and Subendometrial Blood Flow
Acronym: PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mostafa Abdo Ahmed, Principal Investigator, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB#: 2774/11-72016
Record Dates: First submitted 2017-11-02; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Laparoscopic ovarian drilling; subendometrial blood flow
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Intervention Model Description: Laparoscopic ovarian drilling was performed under general anesthesia with good muscle relaxation and endotracheal intubation using the three-punctures technique (one puncture 10mm at the umbilicus and the other two punctures 5mm at both iliac fossa) in the early follicular phase. A specially designed monopolar electrocautery probe was used to penetrate the ovarian capsule at 4 points (regardless of the size of the ovary), with the aid of a short burst of monopolar diathermy. The probe (which has a distal stainless steel needle measuring 10 mm in length and 2 mm in diameter) was applied to the surface of the ovary at a right angle to avoid slippage and to minimize surface damage. A monopolar coagulating current at a 40 W power setting was used. The needle was pushed through the ovarian capsule for about 4 mm depth into the ovarian tissue and electricity was activated for 4 seconds. The ovary was then cooled using 200 ml crystalloid solution before releasing the ligament.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- polycystic ovary syndrome patients (Experimental): patients with polycystic ovary syndrome performed laparoscopic ovarian drilling to induce ovulation
  Interventions: Procedure: Laparoscopic ovarian drilling

INTERVENTIONS:
Procedure: Laparoscopic ovarian drilling — A specially designed monopolar electrocautery probe was used to penetrate the ovarian capsule at 4 points, with the aid of a short burst of monopolar diathermy. The probe (which has a distal stainless steel needle measuring 10 mm in length and 2 mm in diameter) was applied to the surface of the ovary at a right angle to avoid slippage and to minimize surface damage. A monopolar coagulating current at a 40 W power setting was used. The needle was pushed through the ovarian capsule for about 4 mm depth into the ovarian tissue and electricity was activated for 4 seconds.

SUMMARY:
Serum level of total testosterone was measured in the early follicular phase (days 2-4 of spontaneous cycle in oligomenorrhic patients). To start the study in amenorrhic patients (after exclusion of pregnancy) they received progesterone (oral Norethisterone Acetate 10 mg daily for 5 days) to induce withdrawal bleeding and total testosterone was measured in days 2-4 of this withdrawal bleeding.

Color Doppler ultrasound scanning will be performed to assess the subendometrial blood flow. The subendometrial region was observed and analyzed in each woman using color and power Doppler flow ultrasonography. By means of color and power Doppler flow imaging, color signals was searched for in the subendometrial region and areas of maximum color intensity, representing the greatest Doppler frequency shifts, was visualized, then selected for pulsed Doppler examination. Pulsatility index (PI) and resistance index (RI) were calculated in each selected Doppler wave.

Laparoscopic ovarian drilling was performed under general anesthesia with good muscle relaxation and endotracheal intubation using the three-punctures technique (one puncture 10mm at the umbilicus and the other two punctures 5mm at both iliac fossa) in the early follicular phase (after stoppage of menstrual or withdrawal bleeding).

A specially designed monopolar electrocautery probe was used to penetrate the ovarian capsule at 4 points (regardless of the size of the ovary), with the aid of a short burst of monopolar diathermy. The probe (which has a distal stainless steel needle measuring 10 mm in length and 2 mm in diameter) was applied to the surface of the ovary at a right angle to avoid slippage and to minimize surface damage. A monopolar coagulating current at a 40 W power setting was used. The needle was pushed through the ovarian capsule for about 4 mm depth into the ovarian tissue and electricity was activated for 4 seconds. The ovary was then cooled using 200 ml crystalloid solution before releasing the ligament.

Follow up:

Total testosterone and blood flow assessment (PI - RI) of the subendometrial region were performed again in the early follicular phase (days 2-4 of the menstrual cycle) of the first post-operative spontaneous menstruation (which occurred within 10 weeks after the operation).

Also, patients were followed to detect ovulation. ovulating patients were followed for 6 months to detect pregnancy.

DETAILED DESCRIPTION:
Effect of Laparoscopic Ovarian Drilling on Subendometrial Blood Flow in Women with Polycystic Ovary Syndrome

Patients and methods:

This interventional study was carried out in the Department of Obstetrics and Gynecology (Infertility, Ultrasound and Gynecologic endoscopy units), Faculty of Medicine, Zagazig University Hospitals in the period between July 2016 and October 2017. The study included 200 infertile women (primary or secondary infertility) with PCOS attended the infertility outpatient clinic and fulfilled the following inclusion criteria: 1- Patients' ages 20 to 34 years; 2- BMI 18-25 kg/m2; 3- PCOS was diagnosed according to Rotterdam criteria, 2003 (two criteria are sufficient for diagnosis of PCOS): (i) oligo-and/or an-ovulation; which is manifested clinically by amenorrhoea or oligomenorrhoea, (ii) hyperandrogenism (clinical and/or biochemical); (hirsutism and/or elevated serum level of total testosterone), (iii) polycystic ovaries by ultrasound (each ovary contains 12 or more follicles measuring 2-9 mm and/ or ovarian volume more than 10 ml), ( we included only patients who had the three criteria of PCOS) , and previously documented anovulation by transvaginal ultrasound follicular monitoring while taking incremental doses of clomiphene citrate (clomiphene citrate resistant); 4- Hysterosalpingography and husband semen analysis were normal in all subjects. 5- All women in the study were free of any medical illness and had not received any medications in the last 6-9 months before the study apart from clomiphene citrate.

Exclusion criteria were: 1- Other PCOS like syndromes (late onset congenital adrenal hyperplasia-androgen producing tumors-Cushing,s syndrome), hyperprolactinemia and thyroid abnormalities; 2- Gross ovarian pathology either diagnosed preoperatively by ultrasound or intraoperatively by laparoscopy; 3- Any uterine pathology diagnosed preoperatively by ultrasound, HSG or hysteroscopy; or intraoperatively by endoscopy and suspected to cause infertility; 3- Other causes of infertility even if diagnosed during laparoscopy such as tubal pathology and pelvic endometriosis or adhesions; 4- Previous uterine, tubal or ovarian surgery. 5- Contraindications to laparoscopy and general anesthesia; 6- Pregnancy before the first post-operative menstrual cycle.

After full detailed history taking, general, abdominal and local examination and exclusion of any associated medical disorders, transabdominal and/or transvaginal ultrasound was done to exclude patients with ovarian or pelvi-abdominal masses. Other investigations were done to fulfill the inclusion and exclusion criteria (serum prolactin level, free T3, free T4, TSH). Serum level of total testosterone was measured in the early follicular phase (days 2-4 of spontaneous cycle in oligomenorrhic patients). To start the study in amenorrhic patients (after exclusion of pregnancy) they received progesterone (oral Norethisterone Acetate 10 mg daily for 5 days) to induce withdrawal bleeding and total testosterone was measured in days 2-4 of this withdrawal bleeding. Total testosterone was done for all patients in the Laboratory of Zagazig University Hospitals by Electrochemiluminescence (ECL) technology (Cobas e 411 analyzer-Roche Diagnostics GmbH-D-68298 Mannheim-Germany).

Transvaginal 2D color Doppler probe of Voluson 730 pro V machine (GE healthcare, Austria with a 3.5 MHz sector transducer for TAS and 7.5 MHz sector transducer for TVS) was used. While the patients in lithotomy position after evacuation of their urinary bladder and on the same days of total testosterone level assay, baseline 2D TVS was used to examine the uterus for any abnormality and measuring the uterine size and endometrial thickness and then to identify PCO criteria in both ovaries and ovarian volume was measured using ellipisoid prolate formulae (length X width X height X 0.523, which is calculated automatically by the software of the ultrasound machine), (each ovary contains 12 or more follicles measuring 2-9 mm and/ or ovarian volume more than 10 ml) then color Doppler ultrasound scanning will be performed to assess the subendometrial blood flow. The subendometrial region was observed and analyzed in each woman using color and power Doppler flow ultrasonography. By means of color and power Doppler flow imaging, color signals was searched for in the subendometrial region and areas of maximum color intensity, representing the greatest Doppler frequency shifts, was visualized, then selected for pulsed Doppler examination. Pulsatility index (PI) and resistance index (RI) were calculated in each selected Doppler wave.

Laparoscopic ovarian drilling was performed under general anesthesia with good muscle relaxation and endotracheal intubation using the three-punctures technique (one puncture 10mm at the umbilicus and the other two punctures 5mm at both iliac fossa) in the early follicular phase (after stoppage of menstrual or withdrawal bleeding). The zero-degree telescope (Karl Storz, Tuttlingen, Germany) was introduced to visualize the peritoneal cavity. The pelvis was thoroughly inspected for any pathology and the ovaries were examined for the features of polycystic ovary (bilateral ovarian enlargement with smooth glistening surface unbroken by the usual wrinkles and thick, smooth, whitish capsule). Methylene blue test was done for all patients to examine the tubal patency and bilateral tubal patency is mandatory before ovarian drilling.

A specially designed monopolar electrocautery probe was used to penetrate the ovarian capsule at 4 points (regardless of the size of the ovary), with the aid of a short burst of monopolar diathermy. The probe (which has a distal stainless steel needle measuring 10 mm in length and 2 mm in diameter) was applied to the surface of the ovary at a right angle to avoid slippage and to minimize surface damage. A monopolar coagulating current at a 40 W power setting was used. The needle was pushed through the ovarian capsule for about 4 mm depth into the ovarian tissue and electricity was activated for 4 seconds. The ovary was then cooled using 200 ml crystalloid solution before releasing the ligament.

Follow up:

Total testosterone and blood flow assessment (PI - RI) of the subendometrial region were performed again in the early follicular phase (days 2-4 of the menstrual cycle) of the first post-operative spontaneous menstruation (which occurred within 10 weeks after the operation). In non-menstruating patients, total testosterone and the blood flow assessment were performed by the end of the 10 weeks. In menstruating patients, this cycle was monitored to detect ovulation. Ovulation was assessed by serial transvaginal ultrasound until visualization of pre-ovulatory follicle of at least 18 mm. Ovulation was confirmed by seeing follicle collapse on subsequent transvaginal ultrasound, appearance of fluid in the Cul-de-sac and elevated mid-luteal serum progesterone level >5 ng/ml. Ovulating group was informed to report the occurrence of natural conception for 6 months after LOD. Pregnancy was diagnosed by positive pregnancy test with seeing intrauterine gestational sac by transvaginal ultrasound.

Patients who did not menstruate (pregnancy was excluded at first) or did not ovulate within 10 weeks after drilling as evidenced by poor or no follicular growth by serial transvaginal ultrasound folliculometry, and low mid-luteal serum progesterone level < 5 ng/ml were referred to another group of researchers for re-evaluation

ELIGIBILITY:
Inclusion Criteria:

* Patients' ages 20 to 34 years.
* BMI 18-25 kg/m2.
* PCOS was diagnosed according to Rotterdam criteria, 2003 (two criteria are sufficient for diagnosis of PCOS): (i) oligo-and/or an-ovulation; which is manifested clinically by amenorrhoea or oligomenorrhoea, (ii) hyperandrogenism (clinical and/or biochemical); (hirsutism and/or elevated serum level of total testosterone), (iii) polycystic ovaries by ultrasound (each ovary contains 12 or more follicles measuring 2-9 mm and/ or ovarian volume more than 10 ml), ( we included only patients who had the three criteria of PCOS) , and previously documented anovulation by transvaginal ultrasound follicular monitoring while taking incremental doses of clomiphene citrate (clomiphene citrate resistant).
* Hysterosalpingography and husband semen analysis were normal in all subjects.
* All women in the study were free of any medical illness and had not received any medications in the last 6-9 months before the study apart from clomiphene citrate.

Exclusion Criteria:

* Other PCOS like syndromes (late onset congenital adrenal hyperplasia-androgen producing tumors-Cushing,s syndrome), hyperprolactinemia and thyroid abnormalities.
* Gross ovarian pathology either diagnosed preoperatively by ultrasound or intraoperatively by laparoscopy.
* Any uterine pathology diagnosed preoperatively by ultrasound, HSG or hysteroscopy; or intraoperatively by endoscopy and suspected to cause infertility.
* Other causes of infertility even if diagnosed during laparoscopy such as tubal pathology and pelvic endometriosis or adhesions.
* Previous uterine, tubal or ovarian surgery.
* Contraindications to laparoscopy and general anesthesia.
* Pregnancy before the first post-operative menstrual cycle.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Subendometrial blood flow | Within 10 weeks
  change in Subendometrial blood flow after laparoscopic ovarian drilling

SECONDARY OUTCOMES:
Ovulation | Within 10 weeks
  Ovulation was assessed by serial transvaginal ultrasound until visualization of pre-ovulatory follicle of at least 18 mm. Ovulation was confirmed by seeing follicle collapse on subsequent transvaginal ultrasound, appearance of fluid in the Cul-de-sac and elevated mid-luteal serum progesterone level >5 ng/ml.
Pregnancy | Within 6 months
  Ovulating group was informed to report the occurrence of natural conception for 6 months after LOD. Pregnancy was diagnosed by positive pregnancy test with seeing intrauterine gestational sac by transvaginal ultrasound.